CLINICAL TRIAL: NCT01957137
Title: InterStim® Sacral Nerve Modulation Cycling Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1670
Record Dates: First submitted 2013-06-25; First posted 2013-10-08 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Urinary Urge Incontinence
Keywords: Urinary; Urge; Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Continuous (Other): The device parameter will be continuous.
  Interventions: Device: InterStim® (Device Programming)
- Cycling Parameter #1 (Other): The device parameter will be cyclic program #1.
  Interventions: Device: InterStim® (Device Programming)
- Cycling Parameter #2 (Other): The device parameter will be cyclic program #2.
  Interventions: Device: InterStim® (Device Programming)
- Cycling Parameter #3 (Other): The device parameter will be cyclic program #3.
  Interventions: Device: InterStim® (Device Programming)
- No Stimulation (Other): Following the randomized portion of the study, an assessment was conducted to estimate the effect of a month of no stimulation on incontinence.
  Interventions: Device: InterStim® (Device Programming)

INTERVENTIONS:
Device: InterStim® (Device Programming)

SUMMARY:
The study will assess the effects of different InterStim cycling settings on urinary urge incontinence.

DETAILED DESCRIPTION:
This feasibility study will assess the following outcomes:

* Voiding diaries
* Patient reported assessments of response or satisfaction
* Adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Implanted with either Neurostimulator Model 3023 (InterStim) or Neurostimulator Model 3058 (InterStim II) for at least 3 months
2. Implanted with tined lead models 3889 or 3093
3. Tined lead is located at S3 as determined by sensory or motor responses or x-ray or fluoroscopy
4. Currently showing some efficacy with an InterStim device but has the potential to be optimized per the opinion of the Investigator
5. Primary diagnosis before InterStim implant is urinary urge incontinence.
6. Must be willing to maintain her current regimen (dosage and frequency) of any overactive bladder (OAB) medication (anticholinergic, antimuscarinic or Myrbetriq (Mirabegron)) or tricyclic antidepression medication over the study duration, if applicable.
7. Female subject 18 years of age or older
8. Willing and able to accurately complete voiding diaries and questionnaires, attend visits (within the visit windows +7 days), and comply with the study protocol that includes maintenance of InterStim programming settings over the course of the study
9. Have had no more than one (InterStim) reprogramming at or within 28 days at or prior to randomization
10. Able to consent to participate by signing the Informed Consent Form

    Exclusion Criteria:
11. History of Multiple sclerosis
12. History of Reiter's syndrome
13. History of spinal cord injury or a cerebral vascular accident (CVA)
14. History of diabetes unless the diabetes is well-controlled through diet and/or medications
15. Active symptomatic urinary tract infection (UTI)
16. Stress incontinence as the primary diagnosis
17. Urgency frequency as a primary diagnosis
18. Pelvic pain of uncertain etiology that is not associated with a voiding dysfunction or where pelvic pain is the primary diagnosis
19. Interstitial cystitis as the primary diagnosis
20. Urinary retention as the primary diagnosis
21. Treatment of urinary symptoms with botulinum toxin in the past 12 months or any plan to have botulinum toxin treatment during the study
22. Bilateral lead placement
23. Have other implantable neurostimulator, pacemaker, or defibrillator
24. Have knowledge of planned diathermy, microwave exposure, high output ultrasonic exposure, RF energy exposure, or MRI scans not included within the scanning conditions provided within the MRI Guidelines for InterStim Therapy neurostimulation systems.
25. Have an anticipated system modification within the next 5 months
26. Women who are pregnant or planning to become pregnant (women of child-bearing potential must undergo a pregnancy test, with a clear negative result, no more than 7 days prior to randomization visit)
27. Subjects who frequently use the patient programmer to change device program settings ("frequently" is defined as at least once a day and does not include shutting off the device for safety purposes)
28. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol.
29. Study site personnel will contact the Medtronic Study Manager (or designee) to determine if a potential subject who plans to enroll in an investigational device or drug trial, or is currently enrolled in an investigational device or drug trial is eligible for this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven W Siegel, MD, Principal Investigator — Metro Urology; Shaw Zhou, MD, Principal Investigator — Pinellas Urology, Inc.; Karl Kreder, Jr., MD, MBA, Principal Investigator — University of Iowa Healthcare
Locations (3):
- United States (3):
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - University of Iowa Healthcare, Iowa City, Iowa
  - Metro Urology, Woodbury, Minnesota

REFERENCES:
- [Result] Siegel S, Kreder K, Takacs E, McNamara R, Kan F. Prospective Randomized Feasibility Study Assessing the Effect of Cyclic Sacral Neuromodulation on Urinary Urge Incontinence in Women. Female Pelvic Med Reconstr Surg. 2018 Jul/Aug;24(4):267-271. doi: 10.1097/SPV.0000000000000457. PMID 28914707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty subjects were enrolled into the study from Sept 10, 2013 through May 22, 2015 from 3 US centers.
Groups:
- All Study Participants: Thirty subjects were randomized to 1 of 24 sequences with 4 cycling settings: 2 subjects discontinued early with 1 due to an AE, and 1 due to consent withdrawal. Twenty-eight subjects completed the randomization sequences . After that all subjects went through no stimulation for approximately 4 weeks, which was not part of randomization.
Period: Randomized Portion
Arm/Group | All Study Participants
Started | 30
Continuous Stimulation | 29 (Subjects received continuous stimulation for approximately 4 weeks.)
Cycling Parameter #1 | 30 (Subjects received Cycling Parameter #1 for approximately 4 weeks.)
Cycling Parameter #2 | 28 (Subjects received Cycling Parameter #2 for approximately 4 weeks.)
Cycling Parameter #3 | 28 (Subjects received Cycling Parameter #3 for approximately 4 weeks.)
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: No Stimulation
Arm/Group | All Study Participants
Started | 28 (Following randomized portion, all subjects went through no stimulation for approximately 4 weeks.)
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline descriptions provided were based on 24 subjects who first finished their randomized sequences who were included in the primary analysis.
Groups:
- Subjects Who First Finished Unique Randomization Sequences: Baseline descriptions provided were based on 24 subjects who first finished unique randomization sequences, which are those subjects included in the primary analysis of the primary outcome.
Arm/Group | Subjects Who First Finished Unique Randomization Sequences
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — At time of consent
  years | 64.0 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Years implanted with InterStim therapy [Mean (Standard Deviation); unit: years] | 2.8 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Urinary Urge Incontinent (UUI) Episodes Per Day - Randomized Portion
Description: Urinary urge incontinent episodes were collected through a diary on daily basis for approximately 4 weeks when subjects were under each cycling setting. Only the last 7-day diaries were used for the analysis. The first 3 weeks were used as an adjustment period.
Time Frame: 4 weeks
Population: 24 subjects who first completed the unique randomization sequences were included in the analysis.
Measure: Mean (Standard Deviation); unit: Number of UUI episodes/ Day
Groups:
- Continuous: Subjects received continuous stimulation for approximately 4 weeks.
- Cycling Parameter #1: Subjects received cycling parameter #1 for approximately 4 weeks.
- Cycling Parameter #2: Subjects received cycling parameter #2 for approximately 4 weeks.
- Cycling Parameter #3: Subjects received cycling parameter #3 for approximately 4 weeks.
Arm/Group | Continuous | Cycling Parameter #1 | Cycling Parameter #2 | Cycling Parameter #3
Number analyzed (Participants) | 24 | 24 | 24 | 24
Number of UUI episodes/ Day | 1.64 (1.40) | 1.82 (1.97) | 1.44 (1.20) | 1.76 (1.76)
Statistical Analysis 1: Comparison: Continuous vs Cycling Parameter #1 vs Cycling Parameter #2 vs Cycling Parameter #3; Test type: Superiority or Other; p = 0.3773, Mixed Models Analysis; The final model included cycling, period and the interaction between cycling and period

2. Secondary Outcome: Degree of Urgency - Randomized Portion
Description: Each UUI episode was rated on following scales: 0=None, 1=Mild, 2=Moderate, 3=Severe, which were collected through a diary on daily basis for approximately 4 weeks when subjects were under each cycling setting. The average degree of urgency per UUI episode was calculated from the last 7-day diaries were used for the analysis. The first 3 weeks were used as an adjustment period.
Time Frame: 4 week
Population: 24 subjects who first completed unique randomization sequences were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Continuous | Cycling Parameter #1 | Cycling Parameter #2 | Cycling Parameter #3
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | 1.83 [1.48 to 2.19] | 1.80 [1.44 to 2.16] | 1.54 [1.17 to 1.91] | 1.65 [1.29 to 2.01]
Statistical Analysis 1: Comparison: Continuous vs Cycling Parameter #1 vs Cycling Parameter #2 vs Cycling Parameter #3; Test type: Superiority or Other; p = 0.2396, Mixed Models Analysis; The final model included cycling and period

3. Secondary Outcome: Number of Pads Used Per Day - Randomized Portion
Description: Number of pad use were collected through a diary on daily basis for approximately 4 weeks when subjects were under each cycling setting. Only the last 7-day diaries were used for the analysis. The first 3 weeks were used as an adjustment period.
Time Frame: 4 weeks
Population: 24 subjects who first completed unique randomization sequences were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Pads per day
Arm/Group | Continuous | Cycling Parameter #1 | Cycling Parameter #2 | Cycling Parameter #3
Number analyzed (Participants) | 24 | 24 | 24 | 24
Pads per day | 1.10 [0.67 to 1.52] | 1.16 [0.73 to 1.58] | 1.17 [0.74 to 1.59] | 1.20 [0.78 to 1.63]
Statistical Analysis 1: Comparison: Continuous vs Cycling Parameter #1 vs Cycling Parameter #2 vs Cycling Parameter #3; Test type: Superiority or Other; p = 0.8874, Mixed Models Analysis; The final model included cycling and period

4. Secondary Outcome: Global Response Assessment (GRA) - Randomized Portion
Description: Summary statistics of GRA at different cycling settings are provided. The GRA assessed incontinence symptoms as compared to symptoms prior to subject's entry into the study. Subjects were asked how much their incontinence changed since starting the study: markedly worse, moderately worse, mildly worse, same, slightly improved, moderately improved, or markedly improved. The responses to the symptom change were categorized into three levels for the analysis: worse (markedly worse, moderately worse, mildly worse), same (same), better (slightly improved, moderately improved, or markedly improved).
  Percentages of subjects reported worse, same or better under each cycling setting since starting the study are presented.
Time Frame: 4 weeks
Population: 24 subjects who first completed unique randomization sequences were included in the analysis.
Measure: Number; unit: Percent of Subjects
Arm/Group | Continuous | Cycling Parameter #1 | Cycling Parameter #2 | Cycling Parameter #3
Number analyzed (Participants) | 24 | 24 | 24 | 24
Percent of Subjects
  Better | 29 | 38 | 54 | 42
  Same | 25 | 21 | 17 | 38
  Worse | 46 | 42 | 29 | 21

5. Secondary Outcome: Number of UUI Episodes Per Day - no Stimulation
Description: UUI episodes were collected through a diary on daily basis for approximately 4 weeks when subjects were under no stimulation. Only the last 7-day diaries were used for the analysis. The first 3 weeks were used as an adjustment period.
Time Frame: 4 Weeks
Population: 28 subjects who received no stimulation were included in the analysis.
Measure: Mean (Standard Deviation); unit: Number of UUI episodes/ Day
Groups:
- No Stimulation: Following the randomized portion of the study, all subjects went through no stimulation for approximately 4 weeks.
Arm/Group | No Stimulation
Number analyzed (Participants) | 28
Number of UUI episodes/ Day | 1.97 (2.04)

6. Secondary Outcome: Degree of Urgency - no Stimulation
Description: Each UUI episode was rated on following scales: 0=None, 1=Mild, 2=Moderate, 3=Severe, which were collected through a diary on daily basis for approximately 4 weeks when subjects were under no stimulation. The average degree of urgency per UUI episode was calculated from the last 7-day diaries were used for the analysis. The first 3 weeks were used as an adjustment period.
Time Frame: 4 weeks
Population: 28 subjects who received no stimulation were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Stimulation
Number analyzed (Participants) | 28
units on a scale | 1.77 (0.64)

7. Secondary Outcome: Number of Pads Used Per Day - no Stimulation
Description: Number of pad use were collected through a diary on daily basis for approximately 4 weeks when subjects were under no stimulation. Only the last 7-day diaries were used for the analysis. The first 3 weeks were used as an adjustment period.
Time Frame: 4 Weeks
Population: 28 subjects who received no stimulation were included in the analysis.
Measure: Mean (Standard Deviation); unit: Pad use / day
Arm/Group | No Stimulation
Number analyzed (Participants) | 28
Pad use / day | 1.23 (1.22)

8. Secondary Outcome: Global Response Assessment - no Stimulation
Description: Summary of GRA under no stimulation setting is provided. The GRA assessed incontinence symptoms as compared to symptoms prior to subject's entry into the study. Subjects were asked how much their incontinence changed since starting the study: markedly worse, moderately worse, mildly worse, same, slightly improved, moderately improved, or markedly improved. The responses to the symptom change were categorized into three levels for the analysis: worse (markedly worse, moderately worse, mildly worse), same (same), better (slightly improved, moderately improved, or markedly improved).
Time Frame: 4 Weeks
Population: 28 subjects who received no stimulation were included in the analysis.
Measure: Number; unit: Percent of Subjects
Arm/Group | No Stimulation
Number analyzed (Participants) | 28
Percent of Subjects
  Better | 43
  Same | 21
  Worse | 36

9. Secondary Outcome: Adverse Events - no Stimulation
Description: Summary of adverse device effects when subjects were under no stimulation is provided. Percentage of subjects experiencing any type of Adverse Device Effect under no stimulation is presented.
Time Frame: 4 Weeks
Population: 28 subjects who received no stimulation were included in the analysis.
Measure: Number; unit: Percent of Subjects
Arm/Group | No Stimulation
Number analyzed (Participants) | 28
Percent of Subjects | 10.7

ADVERSE EVENTS:
Time Frame: 4 Weeks per period, a total of 4 periods in randomization portion. After randomized portion, each subject was under no stimulation for a period of 4 weeks, which was not part of the randomization.
Groups:
- No Stimulation: Subjects received no stimulation for approximately 4 weeks.
Arm/Group | Continuous | Cycling Parameter #1 | Cycling Parameter #2 | Cycling Parameter #3 | No Stimulation
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/29 | 4/30 | 4/28 | 4/28 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous (N=29) | Cycling Parameter #1 (N=30) | Cycling Parameter #2 (N=28) | Cycling Parameter #3 (N=28) | No Stimulation (N=28)
Device stimulation issue (Surgical and medical procedures) | 1 (1) | 4 (4) | 4 (4) | 4 (4) | 0 (0) — Adverse device effects are presented in this table.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No